CLINICAL TRIAL: NCT06551987
Title: Cognitive Behavioral Therapy for Insomnia vs Brief Behavioral Therapy for Insomnia in Military Personnel With Postconcussive Symptoms Following Mild Traumatic Brain Injury
Brief Title: Behavioral Insomnia Treatment in Mild Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Hope Health Research Institute (Unknown)
Responsible Party: Principal Investigator, Kristi Pruiksma, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000222; TP220139 (Other: Department of Defense)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Insomnia; Mild Traumatic Brain Injury
Keywords: Cognitive Behavioral Therapy for Insomnia; Brief Behavioral Therapy for Insomnia; Insomnia; Mild Traumatic Brain Injury; Active Duty Military Personnel
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Concussion | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia (Active Comparator): 6 weekly, 50-minute sessions delivered individually using in-person or telehealth format by a trained behavioral health provider.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Brief Behavioral Therapy for Insomnia (Active Comparator): 4 weekly, 30-minute sessions delivered individually using in-person or telehealth format by a trained behavioral health provider.
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — 6 weekly, 50-minute sessions delivered individually using in-person or telehealth format by a trained behavioral health provider.
  Arms: Cognitive Behavioral Therapy for Insomnia
Behavioral: Brief Behavioral Therapy for Insomnia — 4 weekly, 30-minute sessions delivered individually using in-person or telehealth format by a trained behavioral health provider.
  Arms: Brief Behavioral Therapy for Insomnia

SUMMARY:
This is a single site, two-armed random controlled trials (RCT) comparing six sessions of Cognitive Behavioral Therapy for Insomnia (CBT-I) with four sessions of Brief Behavioral Therapy for Insomnia (BBT-I) in service members with comorbid insomnia and prolonged postconcussive symptoms present for at least 3 months after Mild Traumatic Brain Injury (mTBI).

DETAILED DESCRIPTION:
The purpose of this study is to identify the optimal behavioral treatment for insomnia in service members with comorbid insomnia and prolonged postconcussive symptoms following Mild Traumatic Brain Injury (mTBI). The study will compare Cognitive Behavioral Therapy for Insomnia (CBT-I) and Brief Behavioral Therapy for Insomnia (BBT-I) and determine the impact of behavioral insomnia treatment on insomnia symptom severity. This study will explore the impact of insomnia treatment on prolonged postconcussive symptoms and blood-based biomarkers. The overall objective is to determine if behavioral insomnia therapy can improve outcomes in service members with prolonged postconcussive symptoms following mTBI.

Both in-person and telehealth treatment formats will be offered to adapt to the service members schedule. The minimum acceptable number of sessions to the interventions in order to have evaluable data will be 4 sessions for CBT-I and 3 sessions for BBT-I. A participant is considered to have completed the study if he or she has completed the baseline assessment, at least 4 sessions for CBT-I and 3 sessions for BBT-I, and the 7-week and 12-week follow-up assessments.

Participants will be seen and treated at the Intrepid Spirit Center and/or the STRONG STAR offices both part of the Carl R. Darnall Army Medical Center (CRDAMC) located on the Fort Cavazos. Active duty service members at least 18 years of age who are seeking clinical care for persisting mTBI symptoms at the Intrepid Spirit Center located on Fort Cavazos. Women will be actively recruited into the study.

ELIGIBILITY:
Inclusion Criteria:

* Active duty U.S. military service members.
* At least 18 years of age.
* Ability to provide informed consent and follow study-related instructions.
* Self-report of a Mild Traumatic Brain Injury (mTBI) at least 3 months prior to enrollment based on self-report.
* At least 2 postconcussive symptoms scored > 2 (moderate) on the Neurobehavioral Symptom Inventory (NSI), with at least 1 of these symptoms from the cognitive domain in addition to the sleep disturbances item.
* Clinically significant chronic insomnia disorder assessed by an independent evaluator using the Structured Clinical Interview for Sleep Disorders-Revised (SCISD-R)_No Split Week Self-Assessment of Sleep Survey (SASS-Y).
* Minimum score of 15 on the Insomnia Severity Index (ISI).
* Plans to be in the area for the next 3 months.
* Stable on psychotropic and hypnotic medications for at least 1 month.
* Stable on continuous positive airway pressure therapy if diagnosed with sleep apnea for at least 1 month.

Exclusion Criteria:

* Moderate TBI (e.g., skull fracture, brain hemorrhage, hematoma) indicated by self-report or medical record.
* Any sleep, medical, or psychiatric disorder requiring urgent treatment (e.g., suicide risk, substance use, insomnia with occupational impairment in high risk professions; very short sleep duration of less than 4 hours on average; bipolar disorder or psychosis) or that otherwise interferes with the completion of the baseline assessment.
* Working night shifts (i.e., duty later than 9:00 pm or before 5:30 am) more than 3 times per month.
* Planned major surgery.
* Pregnancy, assessed by self-report and review of medical record.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline, Treatment, 7 Week Follow-up, 12 Week Follow-up
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the last month. Each item on the ISI is rated on a 5-point Likert scale, ranging from 0 (no problem) to 4 (very severe problem), leading to a total possible score between 0 and 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Neurobehavioral Symptom Inventory (NSI) | Baseline, 7 Week Follow-up, 12 Week Follow-up
  The NSI is a 22-item self-report measure that assesses postconcussive symptoms and classifies them into vestibular, somatic, cognitive, and affective factors, and indicates symptom severity. Respondents rate the severity of each symptom on a scale from 0 (none) to 4 (very severe). Total scores range between 0-88.
NIH Toolbox v3 | Baseline, 7 Week Follow-up
  The NIH Toolbox Cognition Domain measures several aspects of cognitive functioning, including language, episodic memory, executive function, working memory and processing speed. It is a battery administered and automatically scored on the iPad, assessing cognitive function. Higher scores indicate higher levels of functioning compared nationally. A score around 130 suggest superior ability, around 115 suggest above-average fluid cognitive ability, around 100 is average compared with others nationally, around 85 suggests significantly below-average, 70 or below suggests very low functioning.

SECONDARY OUTCOMES:
Dysfunctional Beliefs and Attitudes about Sleep (DBAS) | Baseline, 7 Week Follow-up, 12 Week Follow-up
  Consisting of 18 items the DBAS evaluates the presence of and changes in sleep-related beliefs and attitudes. Sixteen items are rated from 0 "Strongly disagree" to 10 "Strongly agree."
Nightmare Disorder Index (NDI) | Baseline, 7 Week Follow-up, 12 Week Follow-up
  The NDI is a 5-item self-report screening measure intended to evaluate symptoms of nightmare disorder according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-5) diagnostic criteria. NDI questions assess nightmare frequency, characteristics, distress, and impairment, and duration nightmares have been experienced with individual ratings ranging from 0 to 4. The index score is calculated by summing the number of nightmares per week (up to 14), number of nights with nightmares per week (0-7), and the frequency of nightmare-related awakenings (0-4), ratings of the severity of the nightmares (0-6), and the intensity of the nightmares (0-6).
Epworth Sleepiness Scale (ESS) | Baseline, Treatment, 7 Week Follow-up, 12 Week Follow-up
  The ESS is an 8-item self-report measure that assesses the likelihood of falling asleep in various situations. The Scale scores, 0 to 5: Low daytime sleepiness (normal), 6 to 10: High daytime sleepiness (normal), 11 to 12: Mild excessive daytime sleepiness, 13 to 15: Moderate excessive daytime sleepiness, and 16 to 24: Severe excessive daytime sleepiness.
Patient Health Questionnaire (PHQ-9) | Baseline, 7 Week Follow-up, 12 Week Follow-up
  The PHQ-9 assesses the frequency of each of the 9 symptoms of major depressive disorder as defined by the DSM-5. Scoring measures severity of depression, as follows 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, 15-19 is moderately severe depression, 20-27 is severe depression.
Multidimensional Fatigue Inventory (MFI-20) | Baseline, 7 Week Follow-up, 12 Week Follow-up
  The MFI-20 is a 20-item measure designed to index dimensions of fatigue: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. MFI scores range from 20-100 (most severe)
Headache Impact Test (HIT-6) | Baseline, 7 Week Follow-up, 12 Week Follow-up
  The HIT-6 is a 6-item measure of headache disability. Each item uses a 5-point Likert scale with higher scores indicating greater severity. The four headache impact severity categories are little or no impact (49 or less), some impact (50-55), substantial impact (56-59), and severe impact (60-78).
General Anxiety Disorder (GAD-7) | Baseline, 7 Week Follow-up, 12 Week Follow-up
  The GAD-7 is a 7-item measure of anxiety severity and impairment. Items use a Likert-type scale, with higher scores indicating greater severity and impairment. Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Depressive Symptoms Index-Suicidality Subscale (DSI-SS) | Baseline, Treatment, 7 Week Follow-up, 12 Week Follow-up
  The DSI-SS assesses current suicidal ideation. The DSI-SS is a 4-item self-report measure of suicidal ideation that focuses on ideation, plans, perceived control over ideation, and impulses for suicide. Scores on each item range from 0 to 3 (total score range 0-12), with higher scores reflecting greater severity of suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Kristi E Pruiksma, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Carl R. Darnall Army Medical Center, Fort Cavazos, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bramoweth AD, Lederer LG, Youk AO, Germain A, Chinman MJ. Brief Behavioral Treatment for Insomnia vs. Cognitive Behavioral Therapy for Insomnia: Results of a Randomized Noninferiority Clinical Trial Among Veterans. Behav Ther. 2020 Jul;51(4):535-547. doi: 10.1016/j.beth.2020.02.002. Epub 2020 Feb 20. PMID 32586428
- [Background] Pruiksma KE, Hale WJ, Mintz J, Peterson AL, Young-McCaughan S, Wilkerson A, Nicholson K, Dondanville KA, Fina BA, Borah EV, Roache JD, Litz BT, Bryan CJ, Taylor DJ; STRONG STAR Consortium. Predictors of Cognitive Behavioral Therapy for Insomnia (CBTi) Outcomes in Active-Duty U.S. Army Personnel. Behav Ther. 2020 Jul;51(4):522-534. doi: 10.1016/j.beth.2020.02.001. Epub 2020 Feb 14. PMID 32586427
- [Background] Mysliwiec V, Martin JL, Ulmer CS, Chowdhuri S, Brock MS, Spevak C, Sall J. The Management of Chronic Insomnia Disorder and Obstructive Sleep Apnea: Synopsis of the 2019 U.S. Department of Veterans Affairs and U.S. Department of Defense Clinical Practice Guidelines. Ann Intern Med. 2020 Mar 3;172(5):325-336. doi: 10.7326/M19-3575. Epub 2020 Feb 18. PMID 32066145